CLINICAL TRIAL: NCT00310297
Title: A Randomized, Open Label, Two-arm, Cross-over Design Study to Compare the Pharmacodynamics and Pharmacokinetics of Insulin Glulisine and Insulin Lispro in Obese Patients With Type 2 Diabetes.
Brief Title: Insulin Glulisine in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_1505
Record Dates: First submitted 2006-03-02; First posted 2006-04-03 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2008-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin Glulisine

SUMMARY:
Primary objective:

To compare the pharmacodynamics of insulin glulisine and insulin lispro injected subcutaneously before three 500 kcal standard meals during a 12 hour day, in obese subjects with type 2 diabetes.

Secondary objectives:

* To compare the pharmacokinetics of insulin glulisine and insulin lispro in obese subjects with type 2 diabetes, injected subcutaneously before three standard meals during a 12-hour day.
* The safety of insulin glulisine, the relationship of the pharmacodynamics and pharmacokinetics with skin thickness and C-peptide, non-esterified fatty acid, triglyceride and β-hydroxybutyrate levels in these subjects will also be assessed.

ELIGIBILITY:
Inclusion criteria :

* Type 2 diabetes mellitus
* Body mass index (BMI) between 35 and 40 kg/m2
* HbA1c ≤10%
* Plasma C-peptide levels ≥0.1 nmol/L.
* Female subjects have to either be postmenopausal, surgically sterilized, or not pregnant and using approved methods of contraception.

Exclusion criteria :

* Type 1 diabetes mellitus, as defined by the World Health Organization
* Subjects currently taking any insulin
* History of hypoglycaemic unawareness
* Injection site skin thickness < or = 8 mm
* Contra-indications from

  * The medical history and physical examination
  * Laboratory tests (haematology, clinical chemistry, and urinalysis by dipstick)
  * Blood pressure and pulse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma glucose concentration (GLUmax, mmol/L) | During the Study Conduct
Maximum plasma glucose excursion (baseline subtracted glucose concentration, ΔGLUmax, mmol/L) | during the study conduct
Time to GLUmax (Tmax, min) | during the study conduct

SECONDARY OUTCOMES:
Area under the insulin concentration-time curve after injection(μIU.min/mL) | between 0 h and 1 h (AUC0-1h), 0 h and 1.5 h (AUC0-1.5h), 0 h and 2 h (AUC0-2h) and 0 h and 4 h (AUC0-4h)
Maximum concentration (Cmax, μIU/mL) | During the study conduct
Adverse events collection | from the inform consnet signed up to the end of the study
Time to maximum concentration (Tmax, min) | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi